CLINICAL TRIAL: NCT02903654
Title: Prevalence of Heterozygote Mothers for Pompe's Disease Among Mothers Having Delivered in French Guiana
Acronym: DEPIPOMP2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: DEPIPOMP2
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Pompe's Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — filter paper
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational

SUMMARY:
Given the high incidence of Pompe's Disease in French Guiana (100 times higher than in mainland France) the aim is to determine the prevalence of heterozygotes among women having just delivered in French Guiana who accepted that their newborn child enters the depipomp1 study. In these women the specific mutations p.Gly648Ser and p.Arg854X will be sought using PCR in order to calculate the prevalence of these mutations and estimate the risk factors associated with them in order to improve genetic counselling.

ELIGIBILITY:
Inclusion Criteria:

* women having delivered in French Guiana whose child was enroled in the depipomp1 study

Exclusion Criteria:

* refusal to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women having delivered in French Guiana whose child was enrolled in the depipomp1 study
Sampling Method: Non-Probability Sample
Enrollment: 925 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
prevalence of p.Gly648Ser and p.Arg854X | Within 3 days after birth
  number of positive mutations divided by total number of women tested